CLINICAL TRIAL: NCT06675812
Title: Improving Help-seeking Propensity Through a Micro-intervention Targeting Common Concerns Among Individuals With Alcohol Problems: A Randomized Controlled Experiment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Centre for Psychiatry Research, Department of Clinical Neuroscience, Karolinska Institutet, & Stockholm Health Care Services (Unknown); Stockholm Center for Dependency Disorders (Unknown)
Responsible Party: Principal Investigator, Magnus Johansson, Dr, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-04537-01
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Abuse; Harmful Alcohol Use; Hazardous Alcohol Use; Hazardous Drinking; Risky Drinking
Keywords: Help-seeking; Treatment gap; Referral to treatment; Social services; Information intervention; Alcohol; Drinking
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): The participant will receive information on what treatment that is offered in their municipal, how the help-seeking process goes (where they can be anonymous etc), and tailored information regarding the barriers that the participant has stated preventing him or her for seeking help today.
  Interventions: Other: Information intervention
- Referral to municipal care (No Intervention): At the anonymous help service where the intervention will be used, is standard practice to refer the person to the municipal care, if he or she request for more help.

INTERVENTIONS:
Other: Information intervention — The participant will receive information on what treatment that is offered in their municipal, how the help-seeking process goes (where they can be anonymous etc), and tailored information regarding the barriers that the participant has stated preventing him or her for seeking help today.
  Arms: Active group

SUMMARY:
Many people who have risky alcohol use or alcohol dependence do not seek help, often is due to concerns about potential consequences or feelings of shame. At the same time, the prognosis is good for those who do seek help and there are effective treatments available.

This project aims to investigate whether increased information about the process can lower these barriers, and in turn encourage more people to seek help for alcohol-related problems.

DETAILED DESCRIPTION:
In Sweden, 4% suffer from alcohol dependency, and up to one-third of all adults have risky consumption of alcohol. This does not only cause suffering for the individual with the problem, but also for their relatives as well as contribute to significant costs for the Swedish society. Moreover, only a small proportion of those with problematic use or dependence of alcohol actually seek-, and receive help. This can be explained by both internal factors, such as feelings of shame and the belief that "one should be able to overcome dependence on their own," as well as external factors like low availability of appealing interventions.

The addiction care in Sweden is unique in that it is a shared responsibility between the regional health care system and the municipalities' social services. The distribution of responsibilities varies significantly across different parts of Sweden, which means that the interventions available to individuals seeking help vary depending on where they live. Previous research has shown that only about 5% of people with alcohol problems wish to seek help through social services, which suggests that in parts of Sweden where social services are the primary treatment option, fewer people may receive help for their issues.

Also, in a previous study that investigated barriers to seek help at social service, fear of consequences and having the problems documented, was identified as one of the largest barriers, with a suggestion that more transparency on how the social service works would reduce this.

Therefore, this study aims to investigate whether more people with problematic alcohol use and alcohol dependency can be encouraged to seek help from social services if they first receive a micro-intervention addressing common barriers to seeking help from social services. The intervention will be based on results from the study mentioned above, targeting the barriers revealed in the results.

The research project will be integrated as an intervention on the already existing website alcoholhjälpen.se, a site and forum run by Region Stockholm that is directed at people with alcohol problems and their relatives throughout Sweden. All users on alcoholhjälpen are anonymous. A new feature will be introduced here: "What help is available locally for me?", which will serve as the entry point to the study. Pre-measurements, consent, phone numbers and email addresses, and the participant's municipality will be collected, as well as asking the participant what is preventing him or her to seek help today. Then the participant will be randomized into either the intervention or control group. The intervention group will receive the micro-intervention, with both information about what is offered in his or her municipality, as well as information about the barriers that the participant has stated. For instance, if the participant has written that fear of losing custody of his or her child, information about how the process goes, and what rights one has as a parent etc will be presented. The control group will receive a referral to their municipality, saying that this is where they seek help. One month later, follow-ups will be conducted to measure the likelihood that the participant will seek help from social services, which is the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Hazardous alcohol use according to AUDIT-C (a score of 3 or more)

Exclusion Criteria:

* Ongoing care contact at a municipal or regional addiction clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Likelihood of seeking help | Four weeks after recieving the intervention
  This will be formulated approximately like this: "How likely are you to seek help for your alcohol use from the municipality?"
  And the response would be on a VAS scale, where 1 is "Very unlikely" and 10 is "Very likely/already have."

SECONDARY OUTCOMES:
Knowledge of available municipal support | Right after receiving the intervention.
  Assessed by participants' self-reported awareness of the help they can receive from their municipality.
  This will be formulated approximately like this: "How well do you know what kind of help you can receive from your municipality?"
  And the response would be on a VAS scale from 1-10.
Confidence in the help-seeking process | Four weeks after recieving the intervention
  Measured by participants' self-reported confidence in how the process works when seeking help from the municipality.
  This will be formulated approximately like this: "How confident do you feel about the process if you seek help from the municipality?"
  And the response would be on a VAS scale from 1-10.
Concerns about negative consequences | Four weeks after recieving the intervention
  Evaluated through participants self-reported worry about potential negative outcomes from seeking help.
  This will be formulated approximately like this: "How worried are you about negative consequences if you seek help from the municipality?"
  And the response would be on a VAS scale from 1-10.
Concerns about confidentiality | Four weeks after recieving the intervention
  Assessed by participants self-reported concerns about maintaining privacy when seeking help.
  This will be formulated approximately like this: "How concerned are you about privacy or that someone you don't want to know might find out if you seek help from the municipality?"
  And the response would be on a VAS scale from 1-10.
Impact of shame on help-seeking behavior | Four weeks after recieving the intervention
  Measured by how much self-reported shame or embarrassment participants reports preventing them from seeking help
  This will be formulated approximately like this: "How much does shame or feeling embarrassed prevent you from seeking help?"
  And the response would be on a VAS scale from 1-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Alkoholhjälpen, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided